CLINICAL TRIAL: NCT01337479
Title: Long-Term Assessment of Treatment Outcomes With Entecavir and Lamivudine for Chronic Hepatitis B Infection in Patients Who Have Enrolled in Phase III Entecavir Trials
Brief Title: A Phase IIIb: Long-Term Outcomes for Hepatitis B (HepB) Patients in Some Previous Entecavir (ETV) Trials
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Other Study IDs: AI463-049
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants of specific phase III entecavir studies: Those who participated in the specific Phase III entecavir studies as described; all had Hepatitis B infections

SUMMARY:
The purpose of this study is to follow patients treated in entecavir Phase III and rollover studies for safety experience and Hepatitis B virus (HBV)-related complications.

DETAILED DESCRIPTION:
Observational Model: Only subjects who participated in Entecavir Phase III studies AI463022, AI463023, AI463026, and AI463027.

Number of groups/cohorts: 1 (All subjects were observed in the same manner).

ELIGIBILITY:
Inclusion Criteria:

* All subjects who participated in Entecavir Phase III studies AI463022, AI463023, AI463026, and AI463027.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Only subjects who participated in Entecavir Phase III studies AI463022, AI463023, AI463026, and AI463027.
Sampling Method: Non-Probability Sample
Enrollment: 1097 (Actual)
Dates: Start 2003-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who have newly reported hepatitis B-related complications during AI463049 (reported by Phase III treatment groups) | data is collected every 6 months
  defined as follows:
  * Hepatic cirrhosis (Diagnosis requires biopsy or imaging study)
  * Esophageal Varices (Grade 1 or higher on endoscopy or barium swallow)
  * Bleeding esophageal varices
  * Ascites (Present on physical exam or imaging study)
  * Hepatic encephalopathy (≥ Stage 2)
  * Hepatocellular carcinoma
  * Spontaneous bacterial peritonitis
  * Gastric varices
  * Bleeding gastric varices
  * Hepatorenal syndrome

SECONDARY OUTCOMES:
To determine the proportion of subjects who have a HBV Deoxyribonucleic acid (DNA) by Polymerase chain reaction (PCR) of < 300 copies/mL over the AI463049 follow-up period by the phase III treatment group | Every 6 months
To determine the proportion of subjects who have Alanine transaminase (ALT) ≤ 1.0 x Upper limit of normal (ULN) over the AI463049 follow-up period by the phase III treatment group | Every 6 months
To determine the proportion of subjects who were Hepatitis B e antigen (HBeAg) positive at the beginning of Phase III trials who have HBeAg loss or HBe seroconversion over the AI463049 follow-up period by the phase III treatment group | Every 6 months
To determine the number of anti-HBV medications following enrollment in AI463049 by the phase III treatment group | Every 6 months
To determine all cause mortality by the phase III treatment group | Every 6 months
To determine HBV-related mortality by the phase III treatment group | Every 6 months
To determine Non-hepatic malignancies by the phase III treatment group | Every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm